CLINICAL TRIAL: NCT02650947
Title: Effects of Sucralose Consumption on Glucose Metabolism, Incretin and Gut Microbiota in Healthy Adult
Brief Title: Sucralose Effects on Glucose Metabolism and Gut Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Collaborators: The Endocrine Society of Thailand (Other)
Responsible Party: Principal Investigator, Chutintorn Sriphrapradang, Assistant Professor, Ramathibodi Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 09-58-16
Record Dates: First submitted 2016-01-02; First posted 2016-01-08 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: Sucralose; Insulin Secretion; Insulin Sensitivity; Incretin; Gut Microbiota; Food and Eating Behaviour; Healthy Volunteers
MeSH Terms: conditions — Insulin Resistance; Feeding Behavior | interventions — trichlorosucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sucralose (Experimental): Subjects in this group ate capsule filled with sucralose 200 mg for 4 weeks (week 1-4) and measured oral glucose tolerance test (OGTT), acute insulin response (AIR), and gut microbe examination at week 4.
  Interventions: Dietary Supplement: Sucralose
- Placebo (Placebo Comparator): Subjects ate empty capsule (placebo) for 4 weeks (week 1-4) and measured OGTT, AIR, and gut microbe examination at week 4.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Sucralose — Consumption of capsules containing either 200 mg sucralose (equivalent to diet soda 3 cans) per day for four weeks
  Other Names: Trichlorosucrose
  Arms: Sucralose
Dietary Supplement: Placebo — Consumption of empty capsule everyday for 4 weeks
  Arms: Placebo

SUMMARY:
Hypothesis:

1. Long-term consumption of sucralose may effect glucose metabolism, incretin hormone secretion and gut microbiota in healthy adults.
2. Long-term consumption of sucralose may alter food behaviour in healthy adults.

DETAILED DESCRIPTION:
Artificial sweeteners such as sucralose, are among the most widely used food additives worldwide. Artificial sweetener consumption is considered safe and beneficial owing to their low caloric content. However, many emerging evidences showed artificial sweeteners may induce glucose intolerance. The objectives of this study were to determine the effect of sucralose on glycemic response, insulin secretion, insulin sensitivity, incretin response, gut microbiota and food behavior in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers without underlying disease
* Normal oral glucose tolerance test
* Agree to participate by written informed consent

Exclusion Criteria:

* Shift workers
* History of diabetes mellitus or prediabetes (impaired fasting glucose and/or glucose tolerance test)
* Malabsorption problem
* Regular consumption of nonnutritive sweeteners
* Liver impairment (aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3-folds upper normal limit)
* Renal impairment (serum creatinine >1.5 mg/dL)
* Use of medications affecting glucose level such as glucocorticoid, estrogen, androgen
* Pregnant and lactating woman
* Smoking within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The effect of sucralose on insulin secretion | 2 hours
  We will measure plasma insulin concentrations before and at 0, 2, 3, 4, 5, 6, 8, 10 minutes after administered intravenously 50%glucose 0.3 g/kg within 1 minute. All these data collected were used to calculate acute insulin response to glucose.

SECONDARY OUTCOMES:
Glucagon-like peptide-1 secretion | 2 hours
Gut microbiota | 4 weeks
  stool exam, polymerase chain reaction for 16s RNA gene using next generation sequencing
Food record | 4 weeks
The effect of sucralose on insulin sensitivity | 2 hours
  We will measure plasma insulin concentrations during an oral glucose tolerance test.

CONTACTS AND LOCATIONS:
Overall Officials: Chutintorn Sriphrapradang, M.D., Principal Investigator — Ramathibodi Hospital
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided